CLINICAL TRIAL: NCT02629315
Title: Lymph Node Yield After Specimen Fixation With Carnoy's Solution and 10% Neutral Buffered Formaldehyde in Patients With Colorectal Cancer or Gastric Adenocarcinoma Specimens: a Randomized Trial
Brief Title: Carnoy's Solution Versus Formalin in Rectal and Gastric Cancer Specimens Following: a Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: NP458/13
Record Dates: First submitted 2015-12-10; First posted 2015-12-14 (Estimated); Last update posted 2020-07-23 (Actual); Status verified 2020-07

CONDITIONS: Rectal Cancer; Gastric Adenocarcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — Carnoy's solution

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Randomization occurred after surgery, the surgeon was blind during the procedure
Oversight: Data Monitoring Committee: No

ARMS (2):
- 10% neutral buffered formaldehyde (Active Comparator): Specimens will be fixed for 24-48hours in 10% neutral buffered formaldehyde and then dissected for lymph nodes.
  Interventions: Other: 10% neutral buffered formaldehyde
- Carnoy's solution (Experimental): Specimens will be fixed for 24-48hours in Carno'ys solution and then dissected for lymph nodes.
  Interventions: Other: Carnoy's solution

INTERVENTIONS:
Other: Carnoy's solution
  Arms: Carnoy's solution
Other: 10% neutral buffered formaldehyde
  Arms: 10% neutral buffered formaldehyde

SUMMARY:
This study evaluates the number of lymph nodes dissected in specimens following fixation with 10% neutral buffered formaldehyde or Carnoy's solution. Specimens were randomized for fixation in each solution.

DETAILED DESCRIPTION:
Carnoy's solution is a tissue fixative that has alcohol allowing for fat clearing along with tissue fixation. Specimens were randomized after the surgical procedure. The perivisceral fat was removed from the stomach and the lymph node stations disected and then fixed in formalin or carnoy's solution for 24-48h. After dissection the residual fat from the formalin group was re-fixed in carnoy and re-disected.

ELIGIBILITY:
Inclusion Criteria - Rectal Cancer:

* Long course neoadjuvant chemoradiation
* Low anterior resection with total mesorectal excision

Inclusion Criteria - Colon Cancer:

- Rectosigmoidectomy

Inclusion Criteria - Gastric Cancer:

* Gastric adenocarcinoma
* Subtotal gastrectomy
* D2 lymphadenectomy

Exclusion Criteria - Rectal Cancer:

* Previous surgery
* Incomplete neoadjuvant chemoradiation
* Refuse to sign the informed consent
* T4b and/or Multivisceral resection

Exclusion Criteria - Colon Cancer:

* Previous surgery
* Neoadjuvant chemoradiation
* Refuse to sign the informed consent
* T4b and/or Multivisceral resection

Exclusion Criteria - Gastric Cancer:

* Distant metastasis
* Previous upper abdomen radiotherapy
* Previous surgery over stomach or omentum
* Refuse to sign the informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2012-05-10 (Actual); Primary Completion 2014-02-10 (Actual); Study Completion 2014-02-10 (Actual)

PRIMARY OUTCOMES:
Lymph node yield | 10 days - accessed with the pathological report for each specimen
  Primary outcome will be the total number of lymph nodes dissected in each specimen

SECONDARY OUTCOMES:
Dissection duration | 10 days - accessed with the pathological report for each specimen
  Secondary outcome will be measured in minutes, counting from the start to the end of the dissection

REFERENCES:
- [Background] Dias AR, Pereira MA, Mello ES, Zilberstein B, Cecconello I, Ribeiro Junior U. Carnoy's solution increases the number of examined lymph nodes following gastrectomy for adenocarcinoma: a randomized trial. Gastric Cancer. 2016 Jan;19(1):136-42. doi: 10.1007/s10120-014-0443-2. Epub 2014 Nov 20. PMID 25410474
- [Background] Pereira MA, Dias AR, Faraj SF, Cirqueira Cdos S, Tomitao MT, Nahas SC, Ribeiro U Jr, de Mello ES. Carnoy's solution is an adequate tissue fixative for routine surgical pathology, preserving cell morphology and molecular integrity. Histopathology. 2015 Feb;66(3):388-97. doi: 10.1111/his.12532. Epub 2014 Nov 10. PMID 25307771
- [Background] Luz DA, Ribeiro U Jr, Chassot C, Collet E Silva Fde S, Cecconello I, Corbett CE. Carnoy's solution enhances lymph node detection: an anatomical dissection study in cadavers. Histopathology. 2008 Dec;53(6):740-2. doi: 10.1111/j.1365-2559.2008.03148.x. No abstract available. PMID 19076686
- [Background] Duldulao M, Booth C, Denham L, Choi A, Friedman G, Kazanjian K. Alcohol fat clearing increases lymph node yield after surgery for colorectal cancer. Am Surg. 2014 Oct;80(10):1054-8. PMID 25264659
- [Background] Scabini S, Montecucco F, Nencioni A, Zoppoli G, Sartini M, Rimini E, Massobrio A, De Marini L, Poggi A, Boaretto R, Romairone E, Ballestrero A, Ferrando V. The effect of preoperative chemoradiotherapy on lymph nodes harvested in TME for rectal cancer. World J Surg Oncol. 2013 Nov 18;11:292. doi: 10.1186/1477-7819-11-292. PMID 24246069
- [Background] Dias AR, Pereira MA, de Mello ES, Nahas SC, Cecconello I, Ribeiro U Jr. Lymph Node Yield After Neoadjuvant Chemoradiotherapy in Rectal Cancer Specimens: A Randomized Trial Comparing Two Fixatives. Dis Colon Rectum. 2018 Aug;61(8):888-896. doi: 10.1097/DCR.0000000000001097. PMID 29944580
- [Derived] Dias AR, Pereira MA, Mello ES, Cecconello I, Ribeiro-Jr U, Nahas SC. CARNOY'S SOLUTION INCREASES LYMPH NODES COUNT IN COLON CANCER SPECIMENS WHEN COMPARED TO FORMALIN FIXATION: A RANDOMIZED TRIAL. Arq Bras Cir Dig. 2022 Jun 17;35:e1656. doi: 10.1590/0102-672020210002e1656. eCollection 2022. PMID 35730885